CLINICAL TRIAL: NCT06119256
Title: Multicenter, Open Label, Single-arm Exploratory Clinical Study of EBV-TCR-T Cells for EBV Infection After Allogenic HSCT
Brief Title: Clinical Study of EBV-TCR-T Cells for EBV Infection After Allogenic HSCT
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Daihong Liu, Director, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S2022-083-01
Record Dates: First submitted 2023-10-21; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-02

CONDITIONS: EBV Infection After Allogenic HSCT
Keywords: EBV infection; allogenic HSCT
MeSH Terms: conditions — Epstein-Barr Virus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EBV-TCR-T cells (Experimental): Phase 1 trail:
  The patients with EBV infection after HSCT will receive one to three infusions of donor-derived EBV-TCR-T cells, with the escalated dose ranging from 5×10^5/kg to 1×10^6/kg EBV-TCR-T cells per dose.
  Phase 2 trail:
  According to the PK and response data, the dose escalation phase will be carried out.
  Interventions: Biological: EBV-TCR-T cells

INTERVENTIONS:
Biological: EBV-TCR-T cells — The patients with EBV infection after HSCT will receive one to three infusions of donor-derived EBV-TCR-T cells, with the escalated dose ranging from 5×10^5/kg to 1×10^6/kg EBV-TCR-T cells per dose.

SUMMARY:
This is a multi-center, single arm, open-label, phase I study to determine the safety and effectiveness of EBV-TCR-T cell immunotherapy in treating EBV virus infection after allogenic HSCT.

DETAILED DESCRIPTION:
EB virus (EBV) infection after allogeneic hematopoietic stem cell transplantation (HSCT) is common and can be lethal without prompt treatment. In this prospective study, HLA-A*02:01/11:01/24:02-restricted EBV-specific T cell receptor (TCR) will be introduced into the T cells of HSCT donors by ex vivo lentiviral transduction to generate EBV-TCR-T cells. An escalated dose ranging from 3×10^5/kg to 1×10^6/kg of EBV-TCR-T cells will be infused into patients with EBV infection. The safety, efficacy, pharmacokinetics and cytokine levels of allogenic EBV-TCR-T cell therapy will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age 14-75 years, gender unlimited.
* Diagnosed with hematologic malignancies and have undergone allogeneic hematopoietic stem cell transplantation (allo-HSCT), with EBV infection after allo-HSCT.
* Karnofsky Score ≥ 70(age ≥16y) or Lansky Score ≥ 50(age<16y).
* TCR-T cell donor inclusion criteria: 1) Age 8-70 years; 2) Understand and voluntarily sign informed consent and are willing to comply with laboratory tests and other research procedures; 3) ≥ 3/6 HLA match with TCR-T cell recipients enrolled; 4) Lymphocyte count = (0.8~4) × 10^9/L; 5) Have sufficient venous circulation, without any symptoms that do not allow blood cell isolation.

Exclusion Criteria:

* Patients with uncontrolled active aGVHD one day before TCR-T cell infusion.
* Patients with severe kidney disease (Cr > 3×normal value), liver damage (TBIL >2.5×upper limit of normal value, ALT and AST > 3×upper limit of normal value) or heart failure (NYHA heart function grade IV) one week before TCR-T cell infusion.
* Anticipated to take immunosuppressive hormones on the day of TCR-T cell infusion.
* Have other malignancies.
* Have relapsed and uncontrolled hematologic malignancies.
* Serologically positive for HIV-Ab or TAP-ab.
* Pregnant or lactating women.
* Anticipated to have other cell therapies in 4 week post TCR-T cell infusion.
* Participated in any other clinical study of drugs and medical devices before 30 days of enrollment.

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse events | 1 year after EBV-TCR-T treatment
  Percentage of participants with adverse events.

SECONDARY OUTCOMES:
Changes of EBV-DNA copies number | 1 year after EBV-TCR-T treatment
  Quantitative PCR will be used to determine viral copy numbers in peripheral blood.
Persistence of EBV-TCR-T cells | 1 year after EBV-TCR-T treatment
  Quantitative PCR using primers specific for the gene encoding EBV-TCR will be used to determine the number of circulating EBV-TCR-T cells in peripheral blood post infusion.
Dose-limiting toxicity | 28 days after EBV-TCR-T treatment
  Toxic effects considered by the investigators to be related to the EBV-TCR-T
Maximum tolerated dose | 28 days after EBV-TCR-T treatment
  The highest dose of DLT was seen in 1/6 of the subjects
The proportion of EBV-DNA negative patients | 180 days after EBV-TCR-T treatment
  The proportion of patients EBV-DNA negative after EBV-TCR-T treatment
The time to EBV-DNA negative | 180 days after EBV-TCR-T treatment
  The time from the start of therapy to EBV-DNA negative detected
The time to response | 180 days after EBV-TCR-T treatment
  The time from the start of therapy to the time when patients firstly achieve complete remission or partial remission
The duration of response | 1 year after EBV-TCR-T treatment
  The time from the patients firstly achieve complete remission or partial remission to progression of disease
The incidence of EBV-PTLD | 1 year after EBV-TCR-T treatment
  The incidence of EBV-PTLD after EBV-TCR-T treatment
The overall response rate to EBV-TCR-T treatment | 28,90,180,365,730 days after EBV-TCR-T treatment
  The overall response rate to EBV-TCR-T treatment
The complete response rate to EBV-TCR-T treatment | 28,90,180,365, and 730 days after EBV-TCR-T treatment
  The complete response rate to EBV-TCR-T treatment
The incidence of EBV reactivation after EBV-TCR-T treatment | 1 year after EBV-TCR-T treatment
  The incidence of EBV reactivation after EBV-TCR-T treatment
Maximum Plasma Concentration (Cmax) of EBV-TCR-T cells | 28 days after EBV-TCR-T treatment
  Pharmacokinetic (PK) parameters of EBV-TCR-T cells in patients with EBV reactivation
Area under the plasma concentration versus time curve (AUC) of EBV-TCR-T cells | 28 days after EBV-TCR-T treatment
  Pharmacokinetic (PK) parameters of EBV-TCR-T cells in patients with EBV reactivation
Half life time (T1/2) of EBV-TCR-T cells | 28 days after EBV-TCR-T treatment
  Pharmacokinetic (PK) parameters of EBV-TCR-T cells in patients with EBV reactivation
Concentration levels of cytokines | 28 days after EBV-TCR-T treatment
  Concentration levels of cytokines (IL-2, IL-6, IL-10, TNF-α, IFN-γ)
Concentration levels of CRP | 28 days after EBV-TCR-T treatment
  Pharmacokinetics of EBV-TCR-T cells
Concentration levels of ferritin | 28 days after EBV-TCR-T treatment
  Pharmacokinetics of EBV-TCR-T cells

CONTACTS AND LOCATIONS:
Overall Officials: Daihong Liu, Doctor, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China